CLINICAL TRIAL: NCT01760694
Title: Multi-Modality Therapy for Untreated Patients With Resectable or Marginally Resectable Pancreatic Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of enrollment
Sponsor: Southwestern Regional Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SRMC 12-08; IORT Pancreatic (Other: Cancer Treatment Centers of America)
Record Dates: First submitted 2012-12-26; First posted 2013-01-04 (Estimated); Last update posted 2014-08-15 (Estimated); Status verified 2014-08

CONDITIONS: Pancreatic Cancer
Keywords: Pancreatic; Pancreas; Intraoperative Radiation Therapy; Chemotherapy
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Surgical Procedures, Operative; Radiation; Drug Therapy; Oxaliplatin; Irinotecan; Fluorouracil; Leucovorin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Resectable Patients (Experimental): Surgery with Intraoperative Radiation Therapy (IORT). Radiation Therapy within 6-8 weeks after surgery followed by FOLFIRINOX every 2 weeks starting within 12 weeks of surgery
  Interventions: Other: Multi-Modality; IORT, Surgery, Radiation, Chemotherapy
- Marginally Resectable Patients (Experimental): 2-3 cycles of neoadjuvant FOLFIRINOX then restaged, then undergo surgery with Intraoperative Radiation Therapy (IORT) within 2-4 weeks following chemotherapy. Then Radiation Therapy within 6-8 weeks followed by FOLFIRINOX every 2 weeks starting within 12 weeks of surgery for a total of 2-4 cycles
  Interventions: Other: Multi-Modality; IORT, Surgery, Radiation, Chemotherapy

INTERVENTIONS:
Other: Multi-Modality; IORT, Surgery, Radiation, Chemotherapy
  Other Names: Intraoperative Radiation Therapy (IORT); Chemotherapy: FOLFIRINOX, Oxaliplatin, Irinotecan, 5-FU, Leucovorin; Surgery: Resectable or Marginally Resectable

SUMMARY:
To assess the ability of a combination of updated and approved modalities in the treatment of first line pancreatic cancer patients to increase the time to Progression Free Survival

DETAILED DESCRIPTION:
For resectable patient; surgery with Intraoperative Radiation Therapy (IORT). Radiation Therapy within 6-8 weeks after surgery followed by FOLFIRINOX every 2 weeks starting within 12 weeks of surgery.

For marginally resectable patients; the patients will have 2-3 cycles of neoadjuvant chemotherapy of FOLFIRINOX and then restaged, undergo surgery with IORT within 2-4 weeks following chemotherapy. Then radiation therapy starting within 6-8 weeks. Followed by FOLFIRINOX every 2 weeks starting within 12 weeks of surgery for a total of 2-4 cycles.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven Exocrine Adenocarcinoma of the pancreas
* Clinically resectable or marginally resectable disease
* No prior radiation or chemotherapy for carcinoma of the pancreas
* ECOG performance status of 0-1
* Patients must be medically able to undergo surgical resection
* Patients of child bearing potential must follow study specific precautions
* Women that are lactating will not be excluded on the condition that they dispose their breast milk.
* Adequate hematologic and biochemical parameters.

Exclusion Criteria:

* Prior treatment for pancreatic cancer.
* Concurrent investigational treatments.
* Unresectable pancreatic mass.
* Neuroendocrine Histological pancreatic cancer
* Distant Metastatic disease
* Any condition that, in the option of the investigator, would compromise the well being of the patient or anything that would prevent the patient from meeting or performing study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2013-01; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Efficacy - Progression Free Survival | 2 years after last patient enrolled
  Interim analysis at specific time points. Measure disease response by CT scans per standard of care or when clinically indicated.

SECONDARY OUTCOMES:
Safety | 2 years after last patient enrolled
  Interim analysis at certain time points. Measure disease response by CT scans per standard of care or when clinically indicated. Collect adverse events and serious adverse events. Collect quality of life data.

CONTACTS AND LOCATIONS:
Overall Officials: Theodore Pollock, DO, Principal Investigator — Southwestern Regional Medical Center, Inc.
Locations (1):
- Southwestern Regional Medical Center, Inc., Tulsa, Oklahoma, United States

REFERENCES:
- See also: Facility website address — http://cancercenter.com